CLINICAL TRIAL: NCT05804123
Title: Application of LiveSpo Navax® in the Treatment Support of Acute Rhinosinusitis and Acute Otitis Media
Brief Title: LiveSpo Navax® Supports the Treatment of Acute Rhinosinusitis and Otitis Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anabio R&D (Industry)
Collaborators: Thai Binh University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TNLS.2021.03; 872/HĐĐĐ (Other: Thai Binh University of Medicine and Pharmacy)
Record Dates: First submitted 2023-03-07; First posted 2023-04-07 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-03

CONDITIONS: Upper Respiratory Tract Infections
Keywords: Acute rhinosinusitis (ARS); Acute otitis media (AOM); Nasal-spraying probiotics; Adult; Children; Infection bacteria; Cytokines; Immunoglobulin A; Bacillus spores
MeSH Terms: conditions — Respiratory Tract Infections; Otitis Media | interventions — Amoxicillin-Potassium Clavulanate Combination; Tablets; Acetylcysteine; xylometazoline; Cefotaxime; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo Navax® and placebo 0.9% NaCl physiological saline are indistinguishable regarding taste and smell. The color and turbidity of LiveSpo Navax® suspension is unrecognizable to investigators except the PI and analyzer, nurses, patient's parents, and patients due to opaque plastic container.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control - Acute rhinosinusitis (ARS) subgroup (Placebo Comparator): The Control - ARS subgroup receives the routine treatment and uses 0.9% NaCl physiological saline:
  Routine treatment (at the Thai Binh Medical University Hospital) is as follows:
  * Oral-administrative antibiotics: Augmentin (Amoxicillin and Acid Clavulanic).
  * Oral-administrative expectorant: Acetylcysteine
  * Nasal- spraying decongestant: Xylometazoline (Otrivin®)
  Interventions: Drug: 0.9% NaCl physiological saline Nasal-spraying; Drug: Augmentin 500Mg Tablet; Drug: Acetylcysteine; Drug: Xylometazoline Nasal
- Navax - Acute rhinosinusitis (ARS) subgroup (Experimental): Navax - ARS subgroup receives the routine treatment and uses NaCl 0.9% plus B. subtilis and B. clausii at 5 billion Colony Forming Units (CFU)/5 mL (LiveSpo® Navax):
  Routine treatment (at the Thai Binh Medical University Hospital) is as follows:
  * Oral-administrative antibiotics: Augmentin (Amoxicillin and Acid Clavulanic).
  * Oral-administrative expectorant: Acetylcysteine
  * Nasal- spraying decongestant: Xylometazoline (Otrivin®)
  Interventions: Combination Product: LiveSpo Navax®; Drug: Augmentin 500Mg Tablet; Drug: Acetylcysteine; Drug: Xylometazoline Nasal
- Control - ARS accompanied by the AOM (ARS & AOM) subgroup (Placebo Comparator): The Control - ARS & AOM subgroup receives the routine treatment and uses 0.9% NaCl physiological saline:
  Routine treatment (at the Thai Binh Children's Hospital) is as follows:
  * Oral-administrative antibiotics: Augmentin (Amoxicillin and Acid Clavulanic). Or injection or infusion-administrative antibiotics such as Imetoxim (Cefotaxime).
  * Antibiotic ear drops: Ciprofloxacin
  * Nasal- spraying decongestant: Xylometazoline (Otrivin®)
  Interventions: Drug: 0.9% NaCl physiological saline Nasal-spraying; Drug: Augmentin 500Mg Tablet; Drug: Xylometazoline Nasal; Drug: Cefotaxime; Drug: Ciprofloxacin
- Navax - ARS accompanied by the AOM (ARS & AOM) subgroup (Experimental): Navax - ARS & AOM subgroup receives the routine treatment and uses NaCl 0.9% plus B. subtilis and B. clausii at 5 billion CFU/5 mL (LiveSpo® Navax):
  Routine treatment (at the Thai Binh Children's Hospital) is as follows:
  * Oral-administrative antibiotics: Augmentin (Amoxicillin and Acid Clavulanic). Or injection or infusion-administrative antibiotics such as Imetoxim (Cefotaxime).
  * Antibiotic ear drops: Ciprofloxacin
  * Nasal- spraying decongestant: Xylometazoline (Otrivin®)
  Interventions: Combination Product: LiveSpo Navax®; Drug: Augmentin 500Mg Tablet; Drug: Xylometazoline Nasal; Drug: Cefotaxime; Drug: Ciprofloxacin

INTERVENTIONS:
Drug: 0.9% NaCl physiological saline Nasal-spraying — 0.9% NaCl physiological saline is prepared by extracting 5 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B.Braun, Germany, product declaration No. VD-32732-19), and then pouring it into the same opaque plastic spraying 10 mL-bottle that is used for LiveSpo Navax.
  Other Names: Registration number: VD-32723-19
  Arms: Control - ARS accompanied by the AOM (ARS & AOM) subgroup; Control - Acute rhinosinusitis (ARS) subgroup
Combination Product: LiveSpo Navax® — In Vietnam, LiveSpo Navax® is manufactured as a Class-A medical device product (Product declaration No.210001337/PCBA-HN) under manufacturing standards approved by Hanoi Health Department, Ministry of Health, Vietnam (Certificate No YT117-19) and ISO 13485:2016
  Other Names: Registration number: No.210001337/PCBA-HN
  Arms: Navax - ARS accompanied by the AOM (ARS & AOM) subgroup; Navax - Acute rhinosinusitis (ARS) subgroup
Drug: Augmentin 500Mg Tablet — Augmentin (GlaxoSmithKline Pte, product declaration No. VN-20169-16) is an oral antibiotic available in the form of 625 mg tablets, which are prescribed as routine treatment for children and adults, respectively.
  Other Names: Registration number: VN-20169-16
Drug: Acetylcysteine — Acetylcysteine 200 mg (STADA Vietnam, product declaration No. VD-22667-15) is an oral expectorant, which is prescribed as routine treatment for children and adults, respectively.
  Other Names: Registration number: VD-22667-15
  Arms: Control - Acute rhinosinusitis (ARS) subgroup; Navax - Acute rhinosinusitis (ARS) subgroup
Drug: Xylometazoline Nasal — Otrivin (Xylometazoline 0.05%) (Novartis VietNam, product declaration No. VN-15558-12) is a nasal-spraying decongestant, which is prescribed as routine treatment for children and adults, respectively.
  Other Names: Otrivin® 0.05 % with Registration number: VN-15558-12
Drug: Cefotaxime — Imetoxim 1g (Cefotaxime 1g) (Imexpharm Pharmaceutical, product declaration No. VD-26846-17) is an injection or infusion-administrative antibiotic, which is prescribed as routine treatment for children.
  Other Names: Imetoxim 1g with Registration number: VD-26846-17
  Arms: Control - ARS accompanied by the AOM (ARS & AOM) subgroup; Navax - ARS accompanied by the AOM (ARS & AOM) subgroup
Drug: Ciprofloxacin — Ciprofloxacin 0.3% (Vidipha Central Pharmaceutical, product declaration No. VD-15205-11) is an antibiotic ear drop, which is prescribed as routine treatment for children.
  Other Names: Registration number: VD-15205-11
  Arms: Control - ARS accompanied by the AOM (ARS & AOM) subgroup; Navax - ARS accompanied by the AOM (ARS & AOM) subgroup

SUMMARY:
Acute respiratory tract infections (ARTIs), such as acute rhinosinusitis (ARS) and acute otitis media (AOM), are common worldwide and caused by viruses or bacteria entering the body through the mouth and nose. AOM frequently occurs in young children and is caused by bacterial reflux into the middle ear. ARS is a relatively common ARTIs and can occur at many ages. To accurately diagnose disease, careful clinical examination and accurate clinical judgment are required, as making a reasonable treatment regimen with the decision to use antibiotics. Probiotics have long been known to have beneficial effects on the digestive system. Not only limited to the gastrointestinal tract but probiotics are also known for their role in reducing infections in the respiratory system. Recently, the investigators have successfully conducted a clinical trial of nasal-spray Bacillus spore probiotics in children infected with respiratory syncytial virus (RSV), and the data show that the probiotics can rapidly and effectively relieve symptoms of RSV-induced ARTIs while exhibiting strong impacts in reducing viral load and inflammation. Here, the investigators conducted a study that directly spraying probiotics into the nose can effectively support to treatment of both ARS and AOM.

The aim of the study about to evaluate the safety and effectiveness of nasal-spraying probiotics containing spores of Bacillus subtilis and Bacillus clausii in the supportive treatment of patients with ARS and AOM.

Study Population: sample size is 120. Description of Sites: the study is carried out at Thai Binh Medical University Hospital and Thai Binh Children's Hospital.

Description of Study Intervention: 120 eligible patients are divided into 2 groups (n=60/group) including the ARS group and the ARS accompanied by the AOM (ARS & AOM) group. 60 patients in each of the above groups were randomly assigned to two subgroups (n=30/subgroup): Patients in the Control-ARS and Control-ARS & AOM subgroups received the routine treatment and three times per day nasal-spraying 0.9% NaCl physiological saline. In contrast, the patients in the Navax-ARS and Navax-ARS & AOM subgroups received three times per day nasal-spraying LiveSpo Navax® in addition to the same standard of care treatment. The standard treatment regimen is 3-7 days, depending on the severity of the disease when the patient arrives for the exam and the progression of the disease during the treatment period.

Study duration: 18 months

DETAILED DESCRIPTION:
Acute rhinosinusitis (ARS) is an inflammation of the nasal passages and the lining of the sinuses due to an infection. Clinical symptoms and signs of ARS include nasal blockage/obstruction/congestion or runny nose, sneezing, headache, sinus pain (facial pain), and loss of smell. According to statistics in the US, there are about 18-22 million ARS visits to the doctor each year that estimated cost of treatment of up to 11 billion dollars. Up to 28.9 million adults were diagnosed with rhinosinusitis, accounting for 11.6% of the population. In a 5-year statistics at the National Otorhinolaryngology Hospital of Vietnam, rhinosinusitis patients in the working age group from 16 to 50 years old account for 87%. Acute otitis media (AOM) is inflammation of the middle ear mucosa accompanied by effusion into the middle ear due to infection, which may be associated with the presence or absence of perforation of the tympanic membrane. Symptoms of AOM include fever, purulent discharge from the ear canal (ear discharge or otorrhea), earache (rubbing or pulling on the earlobe, tossing or turning, difficulty sleeping or crying), headache, and hearing loss temporary (poor response to sound), vomiting or diarrhea. AOM is children's most common ear disease and a common cause of hearing loss. About 90% of children under two years of age have had at least one episode, and about 80% of preschool children have otitis media. The prevalence is now about 20% at 2 years and 8% at the age of 8 years. Bacteria that cause acute rhinosinusitis and acute otitis media include S. pneumoniae, H. influenzae, M. catarrhalis, and S. aureus... Rhinosinusitis and bacterial otitis media usually require antibiotic treatment; however, inappropriate antibiotic therapy will increase drug resistance and side effects, thereby increasing medical costs. In recent years, the role of probiotics in respiratory diseases has also been mentioned in convincing studies. However, these probiotic products are mainly used orally, with very few products being prepared as nasal spray suspensions. Here, the investigators conducted a study that the direct spray of probiotics into the nose effectively supports treating acute rhinosinusitis and acute otitis media.

The objective was to investigate the symptomatic support treatment effects of the probiotic product LiveSpo Navax® as a liquid-suspension form containing Bacillus spores of safe B. subtilis ANA4 and B. clausii ANA39 strains in children and adults having ARS and children having ARS accompanied by AOM caused by bacteria, investigators evaluation of improved symptom efficacy of LiveSpo Navax® in patients; and measurement of changes in bacterial concentrations, and major cytokine indicators in the nasopharyngeal and ear samples before and after 3 days or 7 days using LiveSpo Navax®.

Methods: A randomized, blind, controlled clinical trial is conducted. The patients or parents of patients must provide the following information: full name, sex, age, address…After informed consent,120 eligible patients are divided into 2 groups (n = 60/group each) including the ARS group and the ARS accompanied by the AOM (ARS & AOM) group. 60 patients with ARS will be randomized into two subgroups (n = 30/subgroup): the control - acute rhinosinusitis subgroup (named Control - ARS subgroup) uses 0.9% NaCl physiological saline and an experimental - acute rhinosinusitis subgroup (called the Navax - ARS subgroup) use the probiotics LiveSpo Navax®. And similarly, 60 children with ARS accompanied by AOM will be randomized into two subgroups (n = 30/subgroup): the control - acute rhinosinusitis accompanied by acute otitis media group (named Control - ARS & AOM group) uses 0.9% NaCl physiological saline and an experimental - acute rhinosinusitis accompanied by acute otitis media group (called the Navax - ARS & AOM group) use the probiotics LiveSpo Navax®. The patient is given a coded spray in the form of a blind sample to ensure the study's objectivity. After the follow-up patient time, nasopharyngeal samples on both ARS and ARS accompanied by AOM groups and ear samples on the ARS accompanied by AOM group will be collected at day 0 and day 3 or/and 7 to evaluate potential reductions in bacteria load and modulation of cytokine, IgA, and the presence of probiotic spores in the patient's the nasopharyngeal and ear samples.

Real-time polymerase chain reaction (Real-time PCR) for detection of microorganisms in nasopharyngeal and ear samples: semi-quantitative assays for measuring changes in bacterial concentrations are conducted by the real-time PCR routine protocol, which has been standardized under International Organization for Standardization 5189:2012 (ISO 15189:2012) criteria and used in Vietnam National Children's Hospital. Detection of B. subtilis ANA4 and B. clausii ANA39 are also conducted by real-time PCR SYBR® Green (SYBR® Green is a dsDNA-binding dye), standardized routinely in Spobiotic Research Center, ANABIO R&D Ltd.

ELISA assays for cytokine levels: pro-inflammatory cytokines levels (pg/mL), including interleukin (IL-6, IL-8) and TNF-alpha, and immunoglobin A (ng/mL) are quantified using an enzyme-linked immunosorbent assay kit (ELISA) according to the manufacturer's instructions. The patients are monitored for symptoms of ARS and AOM at days 0, 3, or/and 7, depending on the degree of compliance with the follow-up re-examination of the outpatients. Doctors observe the patient's health conditions, and their patients of information are filled into medical records. During this study, patients are asked to abstain from the consumption of other probiotics, either via nasal spray or oral administration.

Data collection and statistical analysis: individual medical records are collected, and the patient's information is gathered and systematized. The efficacy of LiveSpo Navax® is evaluated and compared to 0.9% Sodium Chloride (NaCl) physiological saline based on the following clinical and sub-clinical criteria obtained in Navax and Control groups: (i) effective the symptomatic-relieving; (ii) the reduction levels (2^△Ct) of bacteria concentrations.△Ct for target genes is calculated as Ct (threshold cycle of real-time PCR assay) at day 3 or/and 7 - Ct at day 0 while Ct of internal control is adjusted to be equal among all samples; (iii) the reduction levels of IL-6, IL-8, and TNF-alpha cytokines and IgA. The tabular analysis is performed on dichotomous variables using the χ2 test or Fisher's exact test when the expected value of any cell is below five. Continuous variables are compared using the Wilcoxon test, t-test, or the Mann-Whitney test when data are not normally distributed. The correlations among the variables are assessed by Spearman's correlation analysis. Statistical and graphical analyses are performed on GraphPad Prism v8.4.3 software (GraphPad Software, CA, USA). The significance level of all analyses is set at p < 0.05. P-values.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute rhinosinusitis: sudden onset of two or more symptoms, one of which should be either nasal blockage/obstruction/congestion or nasal discharge (anterior/posterior nasal drip); and/or facial pain/pressure; and/or reduction or loss of smell for <12 weeks. In children: sudden onset of two or more of the symptoms: nasal blockage/obstruction/congestion or discolored nasal discharge, or cough (daytime and night-time) for < 12 weeks
* Patients diagnosed with acute rhinosinusitis accompanied by acute otitis media: patients from 6 months to 7 years old, suffer from onset ear discharge not caused by otitis external, the tympanic membrane was ruptured with purulent.
* Patients are hospitalized or treated as outpatients but need periodic re-examination
* Have a complete medical record or medical examination book
* For patients under 18 years old, the patient's parents agreed to participate in the study that was explained and signed the study consent form.
* Patients >18 years old: patients agreed to participate in the study, explained, and signed the study consent form.

Exclusion Criteria:

* The patient did not agree to participate in the study.
* There are not enough medical records or medical examination books.
* The patient moves out of the treatment unit (not for professional reasons).
* The outpatients but no periodic re-examination.
* Patients with congenital deafness, or deafness due to neurological causes: meningitis, obstetric complications, ear poisoning...
* Patients with congenital disease-causing disorders of maxillofacial development and mental and physical retardation.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in percentages of patients with free acute rhinosinusitis symptoms | Day 3 compared to Day 0; Day 7 compared to Day 0
  Changes in percentage (%) of acute rhinosinusitis patients with free acute rhinosinusitis symptoms include nasal blockage/obstruction/congestion or runny nose, sneezing, headache, sinus pain (facial pain), loss of smell
Changes in percentages of patients with free acute otitis media symptoms | Day 3 compared to Day 0
  Changes in percentages (%) of acute otitis media patients with free acute otitis media symptoms include fever, purulent discharge from the ear canal (ear discharge or otorrhea), earache (rubbing or pulling on the earlobe, tossing or turning, difficulty sleeping or crying), headache, and hearing loss temporary (poor response to sound), vomiting or diarrhea.

SECONDARY OUTCOMES:
Changes in infection bacterial concentrations can cause acute rhinosinusitis (ARS) and acute otitis media (AOM) | Day 3 compared to Day 0 and/or Day 7 compared to Day 0
  Changes in infection bacterial (S. pneumoniae, H. influenzae, M. catarrhalis) concentrations in nasopharyngeal samples on both ARS and ARS accompanied by AOM groups and ear samples in the ARS accompanied by AOM group, as indicated by real-time PCR threshold cycle (Ct) values
Changes in cytokines level | Day 3 compared to Day 0 and/or Day 7 compared to Day 0
  Changes in levels of tumor necrosis factor-α (TNF-α) (pg/mL), interleukin-6 (IL-6) (pg/mL), and interleukin-8 (IL-8) (pg/mL)... in nasopharyngeal samples on both ARS and ARS accompanied by AOM groups and ear samples in the ARS accompanied by AOM group
Changes in immunoglobulin A level | Day 3 compared to Day 0 and/or Day 7 compared to Day 0
  Changes in level of immunoglobulin A (IgA) (ng/mL) in nasopharyngeal samples on both ARS and ARS accompanied by AOM groups and ear samples in the ARS accompanied by AOM group

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Khieu Huu, MD.,PhD, Principal Investigator — Thai Binh University of Medicine and Pharmacy; Binh Nguyen Thanh, Assoc. Prof., Principal Investigator — Thai Binh University of Medicine and Pharmacy; Anh Nguyen Thị Vân, Assoc. Prof., Principal Investigator — Anabio R&D Ltd
Locations (1):
- Thai Binh University of Medicine and Pharmacy, Thai Binh Medical University Hospital and Thai Binh Children's Hospital, Thái Bình, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), and clinical study report (CSR). For more information or to submit a request, please contact clinicaltrial.probiotics@gmail.com

REFERENCES:
- [Background] Fekete S, Szabo D, Tamas L, Polony G. [The role of the microbiome in otorhinolaryngology]. Orv Hetil. 2019 Sep;160(39):1533-1541. doi: 10.1556/650.2019.31451. Hungarian. PMID 31544493
- [Background] Yoon YK, Park CS, Kim JW, Hwang K, Lee SY, Kim TH, Park DY, Kim HJ, Kim DY, Lee HJ, Shin HY, You YK, Park DA, Kim SW. Guidelines for the Antibiotic Use in Adults with Acute Upper Respiratory Tract Infections. Infect Chemother. 2017 Dec;49(4):326-352. doi: 10.3947/ic.2017.49.4.326. PMID 29299900
- [Background] Zernotti ME, Pawankar R, Ansotegui I, Badellino H, Croce JS, Hossny E, Ebisawa M, Rosario N, Sanchez Borges M, Zhang Y, Zhang L. Otitis media with effusion and atopy: is there a causal relationship? World Allergy Organ J. 2017 Nov 14;10(1):37. doi: 10.1186/s40413-017-0168-x. eCollection 2017. PMID 29158869
- [Background] Rosenfeld RM, Piccirillo JF, Chandrasekhar SS, Brook I, Ashok Kumar K, Kramper M, Orlandi RR, Palmer JN, Patel ZM, Peters A, Walsh SA, Corrigan MD. Clinical practice guideline (update): adult sinusitis. Otolaryngol Head Neck Surg. 2015 Apr;152(2 Suppl):S1-S39. doi: 10.1177/0194599815572097. PMID 25832968
- [Background] Gwaltney JM Jr, Wiesinger BA, Patrie JT. Acute community-acquired bacterial sinusitis: the value of antimicrobial treatment and the natural history. Clin Infect Dis. 2004 Jan 15;38(2):227-33. doi: 10.1086/380641. Epub 2003 Dec 19. PMID 14699455
- [Background] Song M, Hong HA, Huang JM, Colenutt C, Khang DD, Nguyen TV, Park SM, Shim BS, Song HH, Cheon IS, Jang JE, Choi JA, Choi YK, Stadler K, Cutting SM. Killed Bacillus subtilis spores as a mucosal adjuvant for an H5N1 vaccine. Vaccine. 2012 May 9;30(22):3266-77. doi: 10.1016/j.vaccine.2012.03.016. Epub 2012 Mar 22. PMID 22446640
- [Background] Lefevre M, Racedo SM, Ripert G, Housez B, Cazaubiel M, Maudet C, Justen P, Marteau P, Urdaci MC. Probiotic strain Bacillus subtilis CU1 stimulates immune system of elderly during common infectious disease period: a randomized, double-blind placebo-controlled study. Immun Ageing. 2015 Dec 3;12:24. doi: 10.1186/s12979-015-0051-y. eCollection 2015. PMID 26640504
- [Background] Cutting SM. Bacillus probiotics. Food Microbiol. 2011 Apr;28(2):214-20. doi: 10.1016/j.fm.2010.03.007. Epub 2010 Mar 24. PMID 21315976
- [Background] Piewngam P, Zheng Y, Nguyen TH, Dickey SW, Joo HS, Villaruz AE, Glose KA, Fisher EL, Hunt RL, Li B, Chiou J, Pharkjaksu S, Khongthong S, Cheung GYC, Kiratisin P, Otto M. Pathogen elimination by probiotic Bacillus via signalling interference. Nature. 2018 Oct;562(7728):532-537. doi: 10.1038/s41586-018-0616-y. Epub 2018 Oct 10. PMID 30305736
- [Background] Tran DM, Tran TT, Phung TTB, Bui HT, Nguyen PTT, Vu TT, Ngo NTP, Nguyen MT, Nguyen AH, Nguyen ATV. Nasal-spraying Bacillus spores as an effective symptomatic treatment for children with acute respiratory syncytial virus infection. Sci Rep. 2022 Jul 20;12(1):12402. doi: 10.1038/s41598-022-16136-z. PMID 35858943
- [Derived] Khieu TH, Le DP, Nguyen BT, Ngo BT, Chu HT, Truong DM, Nguyen HM, Nguyen AH, Pham TD, Van Nguyen AT. Alleviating symptoms of paediatric acute rhinosinusitis and acute otitis media with otorrhea using nasal-spraying Bacillus probiotics: a randomized controlled trial. Sci Rep. 2025 Jan 27;15(1):3410. doi: 10.1038/s41598-025-87372-2. PMID 39870748